CLINICAL TRIAL: NCT01212250
Title: A Prospective, Double-blind, Randomized Placebo-controlled Trial of Carvedilol for Pre-primary Prophylaxis of Esophageal Varices in Cirrhosis
Brief Title: Carvedilol for Pre-primary Prophylaxis of Esophageal Varices in Cirrhosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ILBS PHT-003
Record Dates: First submitted 2010-09-07; First posted 2010-09-30 (Estimated); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — Carvedilol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carvedilol (Experimental): Tablet 6.25 mg BD
  Interventions: Drug: carvedilol
- placebo (Placebo Comparator): Placebo tablets 2 BD
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: carvedilol — Carvedilol will be administered orally at a start dose of 3.125 mg twice daily. After 1 week, this will increased if systolic blood pressure does not fall below 90 mm Hg. The patient will receive the maximum tolerated dose of carvedilol with a maximum of 6.25 BD.
  Arms: Carvedilol
Drug: Placebo — The placebo tablets will be identical to the carvedilol tablets. First the patients will receive placebo in the dose of 1 BD. Then depending on his tolerance it will be increased to a maximum of 2 BD.
  Arms: placebo

SUMMARY:
Patients of cirrhosis aged 18 to 75 years who have no esophageal varices will be enrolled. After baseline evaluation, the participants will be randomized to receive either Placebo or Carvedilol 12.5 mg BD. After randomization they will be followed up for one year.

ELIGIBILITY:
Inclusion Criteria:

* Patients of cirrhosis aged 18 to 75 years who have no esophageal or gastric varices.

Exclusion Criteria:

* Any contra-indication to beta-blockers
* Any past EVL or sclerotherapy
* Any past history of surgery for portal hypertension
* Significant cardio or pulmonary co-morbidity
* Any malignancy
* Refusal to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2010-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
the proportions of patients who develop esophageal varices at 1 year in each group. | 1 year

SECONDARY OUTCOMES:
Number of patient dying in a period of one year | 1 year
Number of patients needing discontinuation of therapy due to adverse effects. | 1 year
Reduction in Hepatic Venous Pressure Gradient in both groups | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences (ILBS), New Delhi, National Capital Territory of Delhi, India